CLINICAL TRIAL: NCT03886389
Title: The Effects of Insulin and Insulin-related Characteristics, and Short-Term Low-glycemic and High-glycemic Carbohydrate Intervention on Breast Cancer Biomarkers and Survival
Brief Title: Breast Cancer Diet Intervention Study
Acronym: BCDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Haavard Soiland, Professor PhD, Helse Stavanger HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 59
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Early-stage Breast Cancer; Carbohydrate Engorgement; Proliferation; Insulin Resistance; Estrogen Receptor-positive Breast Cancer
Keywords: Breast Cancer; Estrogen receptor positive; Proliferation; Insulin resistance; PROMs; NMRI; RFS; BCSS
MeSH Terms: conditions — Breast Neoplasms; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: None (Open Label) Primary Purpose: Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate/intervention group (Experimental): Breast cancer patients receive 2 x preoperative carbohydrate loading [PreOP(TM)] before surgery; the 1st dose 18 hours before and 2nd dose 2-4 hours before surgery.
  Interventions: Dietary Supplement: PreOP
- Control group (No Intervention): Breast cancer patients receive standard prep fasting procedure with nil food per os 8-10 hours before surgery, drinking tap water until 2 hours before surgery.

INTERVENTIONS:
Dietary Supplement: PreOP — Mixture of Carbohydrates; standard amount designed for enhanced recovery after surgery (ERAS) i.e. preoperative carbohydrate loading before long standing surgery to enhance recovery.
  Arms: Carbohydrate/intervention group

SUMMARY:
The investigators have already proven that Mitotic Activity Index (MAI)is the most robust measure of proliferation in breast cancer tissue.

The purpose was to study whether 18 and 2-4 hours pre-operative per-oral carbohydrate loading (often given in gastrointestinal surgery i.e. enhanced recovery after surgery=ERAS) influences proliferation in the tumor, serum insulin characteristics, metabolic profile and survival.

DETAILED DESCRIPTION:
It has been postulated that a "Western-style" diet, rich in carbohydrates (especially high glycemic carbohydrates) may have an effect on the incidence of breast cancer, and perhaps also prognosis. This may be mediated through the insulin-related pathways in breast cells which may show insulin-dependent proliferation, which may alter outcome.

Aims:

To study:

1. The inter-patient variation in insulin and insulin-related characteristics in the blood taken just before the operation from breast cancer patients, on a usual pre-operative fasting schedule;
2. The influence of the variation in insulin and insulin-related characteristics on proliferation and other cell biological features in the breast cancers of these patients;
3. Whether 4 and 18-hours pre-operative hyperglycaemic glucose loading (to reduce postoperative insulin resistance) influences proliferation (Mitotic Activity Index (MAI) and other cell biological features in breast cancer*
4. The influence of the short-term effect of a pre-operative low-glycaemic carbohydrate isocaloric diet on proliferation and other cell biological features of the primary breast cancer cells (Low-glycemic isocaloric diet intervention study);
5. Epidemiological risk factors: The correlation between epidemiological risk factors, insulin and insulin-related characteristics, proliferation, cell biological features and other biomarkers in breast cancer patients.
6. Estrogen Receptor positive tumors will be analyses separately.
7. Relapse free survival
8. Breast Cancer Specific Survival.

The Short-term effect of carbohydrates will be assessed in a randomized intervention study, where 30 patients receive oral carbohydrates 18 and 4 hours before surgery and 30 patients receive fasting procedure/water.

Primary Outcome

1. Proliferation in the tumor as measured by MAI.

Secondary Outcomes:

1. Serum insulin characteristics (S-insulin, S- insulin c-peptide, S-IGF and S-IGFBP3) will be measured at various peri-surgical timepoints
2. Changes in metabolic profile* in the tumor and in serum samples
3. Patient Reported Outcome Measures (PROM) on well being
4. Relapse free survival
5. Breast Cancer Specific Survival

   * Metabolic profile assessed by High Resolution Magnetic Resonance Spectroscopy (HR-MRS) in the tumor and in serum samples.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive operable patients in 2009-2010, with a clinical and/or radiologic and/or cytologic diagnosis of primary breast cancer, unless the exclusion criteria apply.

Exclusion Criteria:

1. Non-operable patients (i.e" patients with T3-4 (>5 cm) disease or distant metastases at the time of operation).
2. All patients who refuse to participate.
3. All patients with DCIS, micro-invasive cancer < 2mm diameter or tumors with histologic poor-quality material.
4. Co-morbidity (Insulin dependent Diabetes Mellitus, Cushing syndrome, previous or concurrent cancers except CIN and non-melanomatous skin cancer.
5. Mental inability to participate.
6. Persons allergic to one of the compounds in any of the two diets.

Ages: 25 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is 100 x more frequent in women than in men.
Enrollment: 80 (Actual)
Dates: Start 2009-06-12 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Mitotic Activity Index (MAI) | Trough completion of surgery of all included patients, an average of 1,5 years
  Proliferation in invasive front in tumor

SECONDARY OUTCOMES:
S-Insulin | Analysed in serum samples at 5 time points; At inclusion (day 0), admission (day 10), preoperatively (day 11), postoperatively (day12) and at post operative visit (day 30)
  Secretion of insulin into serum; unit, mIE/L (milli international units pr liter)
Well being after surgery | Day 1,2,3,4,5,6 and 7 after surgery
  Patient Reported Outcome Measures (Questionaire)
High Resolution Magnetic Resonance Spectroscopy (HR-MRS) profiling of specific metabolites | Immediately after surgery: tumor is fresh frozen. High Resolution Magnetic Resonance Spectroscopy (HR-MRS) will be done in the fresh frozen tumor and deep frozen serum samples (=as for insulin characteristics)
  Metabolic profiling in the primary tumor and in the serum samples; measure content of lactate, glycine, choline, fatty acids and lipoproteins
Relapse Free Survival | Until 8 years (97 months of follow up)
  Time from surgery to a relapse (Loco-regional, contralateral and systemic) is experienced
Breast Cancer Specific Survival | 8 years follow-up (97 months of follow up)
  Time from surgery to dead of disease or all other causes of death.
S-insulin c-peptide, | Analysed in serum samples at 5 time points; At inclusion (day 0), admission (day 10), preoperatively (day 11), postoperatively (day12) and at post operative visit (day 30)
  Measure of total insulin secreted; unit, nM (nano molar)
S-IGF1 | Analysed in serum samples at 5 time points; At inclusion (day 0), admission (day 10), preoperatively (day 11), postoperatively (day12) and at post operative visit (day 30)
  Measure of Insulin growth factor type 1; unit, nM (nano molar)
S-IGFBP3 | Analysed in serum samples at 5 time points; At inclusion (day 0), admission (day 10), preoperatively (day 11), postoperatively (day12) and at post operative visit (day 30)
  Measure of Insulin growth factor binding protein 3; unit mg/L (milligram per liter)
PR | Trough completion of surgery of all included patients, an average of 1,5 years
  Expression of Progesteron Receptor in the primary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, PhD, Study Director — Helse Stavanger HF; Stavanger University Hospital

IPD SHARING:
Plan to Share IPD: No
All data will be available to all researches involved in the study included the statistician allocated to the study.

REFERENCES:
- [Background] Baak JP, van Diest PJ, Voorhorst FJ, van der Wall E, Beex LV, Vermorken JB, Janssen EA. Prospective multicenter validation of the independent prognostic value of the mitotic activity index in lymph node-negative breast cancer patients younger than 55 years. J Clin Oncol. 2005 Sep 1;23(25):5993-6001. doi: 10.1200/JCO.2005.05.511. PMID 16135467
- [Background] Baak JP, Gudlaugsson E, Skaland I, Guo LH, Klos J, Lende TH, Soiland H, Janssen EA, Zur Hausen A. Proliferation is the strongest prognosticator in node-negative breast cancer: significance, error sources, alternatives and comparison with molecular prognostic markers. Breast Cancer Res Treat. 2009 May;115(2):241-54. doi: 10.1007/s10549-008-0126-y. Epub 2008 Jul 30. PMID 18665447
- [Derived] Lende TH, Austdal M, Bathen TF, Varhaugvik AE, Skaland I, Gudlaugsson E, Egeland NG, Lunde S, Akslen LA, Jonsdottir K, Janssen EAM, Soiland H, Baak JPA. Metabolic consequences of perioperative oral carbohydrates in breast cancer patients - an explorative study. BMC Cancer. 2019 Dec 4;19(1):1183. doi: 10.1186/s12885-019-6393-7. PMID 31801490
- [Derived] Lende TH, Austdal M, Varhaugvik AE, Skaland I, Gudlaugsson E, Kvaloy JT, Akslen LA, Soiland H, Janssen EAM, Baak JPA. Influence of pre-operative oral carbohydrate loading vs. standard fasting on tumor proliferation and clinical outcome in breast cancer patients horizontal line a randomized trial. BMC Cancer. 2019 Nov 8;19(1):1076. doi: 10.1186/s12885-019-6275-z. PMID 31703648